CLINICAL TRIAL: NCT03940742
Title: A Single Dose Pharmacokinetic Study of Tirzepatide in Subjects With Varying Degrees of Hepatic Impairment
Brief Title: A Study of Tirzepatide in Participants With Impaired Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17102; I8F-MC-GPGQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-06-01

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Normal Hepatic Function (Active Comparator): Participants with normal hepatic function received single subcutaneous dose of 5 milligrams (mg) tirzepatide.
  Interventions: Drug: Tirzepatide
- Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment received single subcutaneous dose of 5 mg tirzepatide.
  Interventions: Drug: Tirzepatide
- Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment received single subcutaneous dose of 5 mg tirzepatide.
  Interventions: Drug: Tirzepatide
- Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment received single subcutaneous dose of 5 mg tirzepatide.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176

SUMMARY:
The purpose of this study is to assess how fast tirzepatide gets into the blood stream and how long it takes the body to remove it in participants with impaired liver function compared to healthy participants. The study will last about two months and will include five visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Women of childbearing potential are excluded from the study.
* Women not of childbearing potential may participate and include those who are infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as mullerian agenesis; or postmenopausal
* Are between the body mass index (BMI) of 19.0 and 40.0 kilograms per meter squared (kg/m²), inclusive, at screening

Healthy Participants:

- Healthy males or females as determined by medical history, physical examination, and other screening procedures, with normal liver function

Participants with Impaired Liver Function:

* Males or females with chronic mild, moderate and severe liver impairment, assessed by Child-Pugh scoring
* Have type 2 diabetes mellitus (T2DM) controlled with diet or exercise alone or on stable doses of metformin for at least 8 weeks
* Have a hemoglobin A1c (HbA1c) ≥6.0% and ≤11.0% at screening

Exclusion Criteria:

All Participants:

* Have known allergies to tirzepatide or related compounds
* Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis), elevation in serum amylase or lipase or GI disorder (eg, relevant esophageal reflux or gall bladder disease) or any GI disease which impacts gastric emptying (eg, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by glucagon-like peptide-1 (GLP-1) analogs or dipeptidyl peptidase IV (DPP-IV) inhibitors

Participants with Impaired Liver Function:

* Have hemoglobin <8.5 grams per deciliter (g/dL)
* Have kidney function that is significantly impaired at screening
* Have taken any glucose-lowering medications other than metformin, including insulin, in the past 3 months before screening
* Have brain function impaired significantly due to liver condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Orange County Research Center, Tustin, California
  - Orlando Clinical Research Center, Orlando, Florida
  - New Orleans Center for Clinical Research, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Urva S, Quinlan T, Landry J, Ma X, Martin JA, Benson CT. Effects of Hepatic Impairment on the Pharmacokinetics of the Dual GIP and GLP-1 Receptor Agonist Tirzepatide. Clin Pharmacokinet. 2022 Jul;61(7):1057-1067. doi: 10.1007/s40262-022-01140-3. Epub 2022 Jun 8. PMID 35674880
- See also: A Study of Tirzepatide in Participants With Impaired Liver Function — https://trials.lillytrialguide.com/en-US/trial/3Q0iEn37gojINvezSaoRkX

RESULTS

PARTICIPANT FLOW:
Groups:
- Control (Normal Hepatic Function): Participants with normal hepatic function received single subcutaneous dose of 5 mg tirzepatide.
Period: Overall Study
Arm/Group | Control (Normal Hepatic Function) | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Started | 13 | 6 | 6 | 7
Received at Least One Dose of Study Drug | 13 | 6 | 6 | 7
Completed | 13 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Normal Hepatic Function) | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Total
Number analyzed (Participants) | 13 | 6 | 6 | 7 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (11.3) | 63.2 (4.5) | 51.3 (15.4) | 60.4 (6.6) | 57.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 2 | 8
  Male | 10 | 4 | 5 | 5 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 0 | 4
  Not Hispanic or Latino | 11 | 5 | 5 | 7 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 0 | 3
  White | 11 | 4 | 6 | 7 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 6 | 6 | 7 | 32

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under The Drug Concentration-Time Curve From Zero To Infinity (AUC[0-∞]) of Tirzepatide
Description: Pharmacokinetics (PK): Area Under The Drug Concentration-Time Curve From Zero To Infinity (AUC[0-∞]) of Tirzepatide.
Time Frame: Predose, 8, 12, 24, 48, 72, 96, 168 and 336 post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Control (Normal Hepatic Function) | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 13 | 6 | 6 | 6
nanogram*hour per milliliter (ng*h/mL) | 84300 (28) | 102000 (16) | 82000 (29) | 77000 (33)
Statistical Analysis 1: Comparison: Control (Normal Hepatic Function) vs Mild Hepatic Impairment; Test type: Other; Ratio of geometric least squares mean = 1.08, 90% CI 2-sided [0.879 to 1.32]
Statistical Analysis 2: Comparison: Control (Normal Hepatic Function) vs Moderate Hepatic Impairment; Test type: Other; Ratio of geometric least squares mean = 0.960, 90% CI 2-sided [0.790 to 1.17]
Statistical Analysis 3: Comparison: Control (Normal Hepatic Function) vs Severe Hepatic Impairment; Test type: Other; Ratio of geometric least squares mean = 0.852, 90% CI 2-sided [0.699 to 1.04]

2. Primary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of Tirzepatide
Description: PK: Maximum Observed Drug Concentration (Cmax) of Tirzepatide.
Time Frame: Predose, 8, 12, 24, 48, 72, 96, 168 and 336 post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Control (Normal Hepatic Function) | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 13 | 6 | 6 | 7
ng/mL | 510 (28) | 509 (18) | 516 (44) | 521 (23)
Statistical Analysis 1: Comparison: Control (Normal Hepatic Function) vs Mild Hepatic Impairment; Test type: Other; Ratio of geometric least squares mean = 0.916, 90% CI 2-sided [0.726 to 1.16]
Statistical Analysis 2: Comparison: Control (Normal Hepatic Function) vs Moderate Hepatic Impairment; Test type: Other; Ratio of geometric least squares mean = 1.00, 90% CI 2-sided [0.802 to 1.25]
Statistical Analysis 3: Comparison: Control (Normal Hepatic Function) vs Severe Hepatic Impairment; Test type: Other; Ratio of geometric least squares mean = 0.972, 90% CI 2-sided [0.784 to 1.21]

ADVERSE EVENTS:
Time Frame: Baseline to Study Completion (Up to 14 Months)
Description: All participants who received at least one dose of study drug.
Arm/Group | Control (Normal Hepatic Function) | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6 | 0/6 | 1/7
Other Adverse Events (participants affected / at risk) | 4/13 | 2/6 | 2/6 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Normal Hepatic Function) (N=13) | Mild Hepatic Impairment (N=6) | Moderate Hepatic Impairment (N=6) | Severe Hepatic Impairment (N=7)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Normal Hepatic Function) (N=13) | Mild Hepatic Impairment (N=6) | Moderate Hepatic Impairment (N=6) | Severe Hepatic Impairment (N=7)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT03940742/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT03940742/SAP_001.pdf